CLINICAL TRIAL: NCT00168493
Title: The Neurobiology of Depressive Illness: Causes and Consequences of Altered Brain Monoaminergic Function
Brief Title: The Neurobiology of Depressive Illness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baker Heart Research Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Dr David Barton, Baker Heart Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHMRC D-01
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Major Depression
Keywords: Major Depression; Cardiac disease
MeSH Terms: conditions — Depressive Disorder, Major; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intervention (Active Comparator): there is no sham or placebo control arm It is a single arm study
  Interventions: Drug: antidepressants primarily selective serotonin reuptake inhibitors

INTERVENTIONS:
Drug: antidepressants primarily selective serotonin reuptake inhibitors — normal clinical dosages used according to clinical response as determined by a psychiatrist

SUMMARY:
We aim to determine why patients with depression are at an elevated risk for the development of coronary heart disease, and resolve whether the severity of a patient's depression has a counterpart in demonstrable abnormalities in brain chemistry. Studies will be completed in 28 patients with depression; both males and females. Patients will be studied both untreated and during administration of a selective serotonin re-uptake inhibitor (SSRI) antidepressant. They will be either newly diagnosed with depression, untreated patients suffering a recent relapse, or patients seeking to switch from a non-SSRI antidepressant due to non-response. The turnover of chemical messengers in the brain will be estimated by high internal jugular venous blood sampling and DNA will be isolated and examined from blood cells. Immune function will also be assessed. Whole body and cardiac sympathetic nervous activity will be determined, as well as microneurographic recording of muscle sympathetic nervous activity.

It is hypothesised that patients with depression and no existing demonstrable cardiac disease demonstrate:

Alterations in brain monoaminergic neurotransmitter turnover, resulting in sympathetic nervous activation and dysregulation of the baroreflex control to both the heart (vagal) and muscle vasoconstrictor sympathetic nerves; and Exhibit enhanced platelet reactivity predisposing them to thrombogenesis and myocardial ischaemia.

Therapeutic intervention with an SSRI will modify cardiac sympathetic function, baroreflex sensitivity or platelet reactivity in a fashion likely to reduce cardiac risk.

ELIGIBILITY:
Inclusion Criteria:

* Major depression

Exclusion Criteria:

* heart disease diabetes hypertension psychosis significant suicidal risk dementia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2000-06; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
level of sympathetic nervous system activity and its response to treatment | 12 weeks

SECONDARY OUTCOMES:
clinical response to treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murray A Esler, MBBS Phd, Principal Investigator — Baker Heart Research Insitute
Locations (1):
- Baker Heart Research Institute, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Keating C, Dawood T, Barton DA, Lambert GW, Tilbrook AJ. Effects of selective serotonin reuptake inhibitor treatment on plasma oxytocin and cortisol in major depressive disorder. BMC Psychiatry. 2013 Apr 29;13:124. doi: 10.1186/1471-244X-13-124. PMID 23627666